CLINICAL TRIAL: NCT00336700
Title: A Phase II Study of Gemcitabine and Erlotinib As Adjuvant Therapy In Patients With Resected Pancreatic Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study published November 2010 and no further work will be done
Sponsor: Herbert J. Zeh, III MD, FACS (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Herbert J. Zeh, III MD, FACS, Principal Investigator, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06-016
Record Dates: First submitted 2006-06-12; First posted 2006-06-14 (Estimated); Results first posted 2016-09-19 (Estimated); Last update posted 2016-09-19 (Estimated); Status verified 2016-07

CONDITIONS: Pancreatic Cancer
Keywords: Pancreas; Cancer; Pancreatic
MeSH Terms: conditions — Pancreatic Neoplasms; Neoplasms | interventions — Gemcitabine; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Gemcitabine and Erlotinib (Experimental): Erlotinib (oral) 150 mg/day x 12 months Gemcitabine 1500 mg/m2 IV over 150 minutes q 2 weeks x 4 months
  Interventions: Drug: Gemcitabine; Drug: Erlotinib

INTERVENTIONS:
Drug: Gemcitabine — 1500mg/m2 IV over 150 min IV q 2 weeks 4 months
  Other Names: Gemzar
Drug: Erlotinib — 150 mg/d Daily, oral 12 months
  Other Names: Tarceva

SUMMARY:
Study Hypothesis: To estimate time to recurrence in pancreatic cancer patients treated with adjuvant erlotinib and gemcitabine. Combination therapy will be given for 4 months followed by single agent erlotinib for a total of 12 months.

DETAILED DESCRIPTION:
PATIENT POPULATION Resected pancreatic cancer patients (R0 resection) within 10 weeks of surgery will be eligible, provided that they meet standard eligibility criteria.

STUDY DESIGN Phase II, open-label trial of erlotinib and gemcitabine. SAFETY PLAN Safety as assessed by CTCAE 3.0 STUDY TREATMENT Erlotinib 150 mg/day x 12 months. (oral) Gemcitabine 1500 mg/m2 IV over 150 minutes q 2 weeks x 4 months Patients will be monitored with serial CT scans for the first 2 years after completion of therapy.

Clinical Practice: Therapy will be administered as an outpatient. Primary Evaluations: Time to recurrence CONCOMITANT THERAPY AND CLINICAL PRACTICE No other anti-cancer therapy will be allowed while on study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with potentially resectable pancreatic cancer (including ampullary cancer), prior to or after surgery will be accrued to this study.
* Patients who sign consent prior to surgery must have appropriate diagnostic imaging and be evaluated by one of the surgical co-investigators as having resectable disease, and probable pancreatic adenocarcinoma.
* Patients, who sign consent after surgery, must have adenocarcinoma of the pancreas with negative surgical margins.
* Adjuvant therapy should start within 10 weeks of surgery
* Age 18 years or older
* ECOG performance status of 0 - 1 (see Appendix A)
* Ability to take oral medications without difficulty
* Adequate bone marrow function as evidenced by an absolute neutrophil content (ANC) > 1500/mL and platelet count > 100,000/mL
* Adequate renal function as evidenced by serum creatinine within institutional limits or creatinine clearance > 50 ml/minute if above upper institutional limits (ULN)
* Adequate hepatic function as evidenced by ALT and total bilirubin within 2 times ULN.
* Provision of written informed consent.
* Men and women of childbearing potential must be willing to practice acceptable methods of birth control to prevent pregnancy.

Exclusion Criteria:

* Positive margins on post operative surgical specimen or evidence of metastatic disease (positive retroperitoneal margin is allowed)
* Biliary tree cancers are not allowed (Note: Ampullary cancer allowed).
* Known severe hypersensitivity to erlotinib or any of the excipients of these products
* Any prior treatment with radiation therapy or chemotherapy or vaccines for pancreatic cancer.
* Other coexisting malignancies or malignancies diagnosed within the last 3 years, with the exception of basal cell carcinoma or squamous cell carcinoma of the skin or cervical cancer in situ.
* Concomitant use of phenytoin, carbamazepine, barbiturates, rifampicin, phenobarbital, or St. John's Wort. Other agents which inhibit CYP3A4 may be used with caution (Appendix B)
* Treatment with a non-approved or investigational drug prior to treatment.
* Incomplete healing from previous oncologic or other major surgery.
* Pregnancy or breast feeding (women of childbearing potential).
* As judged by the investigator, any evidence of severe or uncontrolled systemic disease (e.g., unstable or uncompensated respiratory, cardiac, hepatic, or renal disease).
* Evidence of any other significant clinical disorder or laboratory finding that makes it undesirable for the subject to participate in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2006-06; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Herb Zeh, M.D., Principal Investigator — University of Pittsburgh
Locations (1):
- UPMC Cancer Centers Network, Pittsburgh, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Gemcitabine (900-1500 mg/m2) + Erlotinib (50-150 mg Daily): Patients with adenocarcinoma of the pancreas who adjuvant biweekly fixed-dose rate gemcitabine (1500 mg/m2) and daily erlotinib (150 mg/day) for 4 months followed by maintenance erlotinib (150 mg/day) over 8 months.
Period: Overall Study
Arm/Group | Gemcitabine (900-1500 mg/m2) + Erlotinib (50-150 mg Daily)
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Gemcitabine (900-1500 mg/m2) + Erlotinib (50-150 mg Daily)
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 66 [34 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 9

OUTCOME MEASURES:

1. Primary Outcome: Recurrence Free Survival (RFS)
Description: The time interval between day 1, cycle 1, of adjuvant treatment to the first date of radiologic recurrence or death.
Time Frame: Up to 60 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Gemcitabine (900-1500 mg/m^2) + Erlotinib (50-150 mg Daily): Patients with adenocarcinoma of the pancreas who adjuvant biweekly fixed-dose rate gemcitabine (1500 mg/m2) and daily erlotinib (150 mg/day) for 4 months followed by maintenance erlotinib (150 mg/day) over 8 months.
Arm/Group | Gemcitabine (900-1500 mg/m^2) + Erlotinib (50-150 mg Daily)
Number analyzed (Participants) | 25
months | 14 [8.2 to 24.5]

2. Primary Outcome: 1-year Recurrence Free Survival (RFS)
Time Frame: Up to 60 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemcitabine (900-1500 mg/m^2) + Erlotinib (50-150 mg Daily)
Number analyzed (Participants) | 25
percentage of participants | 56 [35 to 73]

3. Primary Outcome: 2-year Recurrence Free Survival (RFS)
Time Frame: Up to 60 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemcitabine (900-1500 mg/m^2) + Erlotinib (50-150 mg Daily)
Number analyzed (Participants) | 25
percentage of participants | 26 [6 to 52]

4. Secondary Outcome: Estimated 1&2 Year Overall Survival (OS)
Description: Time from from date of first study therapy to to death from any cause.
Time Frame: Up to 60 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Gemcitabine (900-1500 mg/m^2) + Erlotinib (50-150 mg Daily)
Number analyzed (Participants) | 25
percentage of participants
  Estimated 1-year OS | 84 [63 to 94]
  Estimated 2-year OS | 53 [22 to 76]

5. Secondary Outcome: Percentage of Participants With Expression of Epidermal Growth Factor Receptor (EGFR)
Description: Percentage of participants with expression of epidermal growth factor receptor (EGFR) expression in the resected tumors was assessed by fluorescence in situ hybridization (FISH) and immunohistochemistry (IHC).
Time Frame: Up to 60 months
Measure: Number; unit: percentage of participants
Arm/Group | Gemcitabine (900-1500 mg/m^2) + Erlotinib (50-150 mg Daily)
Number analyzed (Participants) | 25
percentage of participants
  EGFR FISH - Negative | 80
  EGFR FISH - Positive | 20
  EGFR IHC - 1+ (incomplete circumferential) | 22
  2+ (complete circumferential) | 35
  3+ (complete strong circumferential) | 43

6. Secondary Outcome: KRAS Mutational Status
Description: KRAS mutation status in resected tumor specimens.
Time Frame: Up to 60 months
Measure: Number; unit: percentage of participants
Arm/Group | Gemcitabine (900-1500 mg/m^2) + Erlotinib (50-150 mg Daily)
Number analyzed (Participants) | 25
percentage of participants | 92

ADVERSE EVENTS:
Arm/Group | Gemcitabine (900-1500 mg/m^2) + Erlotinib (50-150 mg Daily)
Serious Adverse Events (participants affected / at risk) | 8/25
Other Adverse Events (participants affected / at risk) | 25/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine (900-1500 mg/m^2) + Erlotinib (50-150 mg Daily) (N=25)
Blood/bone marrow (Blood and lymphatic system disorders) | 3
Gastrointestinal (Gastrointestinal disorders) | 2
Constitutional symptoms (General disorders) | 1
Allergy/immunology (Immune system disorders) | 1
Infection (Infections and infestations) | 4
Musculoskeletal/soft tissue (Musculoskeletal and connective tissue disorders) | 2
Pain (Musculoskeletal and connective tissue disorders) | 1
Dermatology/skin (Skin and subcutaneous tissue disorders) | 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Gemcitabine (900-1500 mg/m^2) + Erlotinib (50-150 mg Daily) (N=25)
Hemoglobin (Blood and lymphatic system disorders) | 10
Dry eye syndrome (Eye disorders) | 2
Ocular/Visual - Other (Eye disorders) | 3
Constipation (Gastrointestinal disorders) | 2
Mucositis/stomatitis (functional/symptomatic), Oral cavity (Gastrointestinal disorders) | 2
Pain, Abdomen NOS (Gastrointestinal disorders) | 3
Mucositis/stomatitis (clinical exam), Oral cavity (Gastrointestinal disorders) | 4
Taste alteration (dysgeusia) (Gastrointestinal disorders) | 4
Vomiting (Gastrointestinal disorders) | 8
Nausea (Gastrointestinal disorders) | 9
Diarrhea (Gastrointestinal disorders) | 18
Constitutional Symptoms - Other (General disorders) | 2
Rigors/chills (General disorders) | 2
Fever (in the absence of neutropenia, where neutropenia is defined as ANC <1.0 x 10^9/L) (General disorders) | 7
Weight loss (General disorders) | 9
Fatigue (asthenia, lethargy, malaise) (General disorders) | 17
Infection - Other (Infections and infestations) | 2
Infection with unknown ANC, Urinary tract NOS (Infections and infestations) | 2
Neutrophils/granulocytes (ANC/AGC) (Investigations) | 3
Bilirubin (hyperbilirubinemia) (Investigations) | 4
Alkaline phosphatase (Investigations) | 5
AST, SGOT(serum glutamic oxaloacetic transaminase) (Investigations) | 6
Leukocytes (total WBC) (Investigations) | 6
ALT, SGPT (serum glutamic pyruvic transaminase) (Investigations) | 7
Dehydration (Metabolism and nutrition disorders) | 2
Calcium, serum-low (hypocalcemia) (Metabolism and nutrition disorders) | 3
Glucose, serum-low (hypoglycemia) (Metabolism and nutrition disorders) | 3
Albumin, serum-low (hypoalbuminemia) (Metabolism and nutrition disorders) | 4
Potassium, serum-low (hypokalemia) (Metabolism and nutrition disorders) | 4
Magnesium, serum-low (hypomagnesemia) (Metabolism and nutrition disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 7
Glucose, serum-high (hyperglycemia) (Metabolism and nutrition disorders) | 11
Joint-function (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness, generalized or specific area (not due to neuropathy), Extraocular (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal/Soft Tissue - Other (Musculoskeletal and connective tissue disorders) | 3
Pain, Back (Musculoskeletal and connective tissue disorders) | 3
Dizziness (Nervous system disorders) | 3
Pain, Head/headache (Nervous system disorders) | 4
Mood alteration, Anxiety (Psychiatric disorders) | 2
Mood alteration, Depression (Psychiatric disorders) | 2
Insomnia (Psychiatric disorders) | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary/Upper Respiratory - Other (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 3
Pruritus/itching (Skin and subcutaneous tissue disorders) | 3
Rash: dermatitis associated with radiation, Chemoradiation (Skin and subcutaneous tissue disorders) | 3
Rash: hand-foot skin reaction (Skin and subcutaneous tissue disorders) | 4
Rash/desquamation (Skin and subcutaneous tissue disorders) | 6
Hair loss/alopecia (scalp or body) (Skin and subcutaneous tissue disorders) | 9
Rash: acne/acneiform (Skin and subcutaneous tissue disorders) | 12
Hypotension (Vascular disorders) | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes